CLINICAL TRIAL: NCT02464345
Title: A Randomised Controlled Trial of a New Integrated Approach to Management of Eating and Weight Disorders, Namely a Healthy APproach to weIght Management and Food in Eating Disorders Compared to Cognitive Behaviour Therapy Enhanced.
Brief Title: Healthy Approach to weIght Management and Food in Eating Disorders (HAPIFED)
Acronym: HAPIFED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: University of Western Sydney (Other)
Responsible Party: Principal Investigator, ANGELICA CLAUDINO, Professor of Psychiatry, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 88881.068180/2014-01
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2019-07

CONDITIONS: Binge Eating Disorder; Bulimia Nervosa; Eating Disorder
Keywords: BED; Binge Eating Disorer; BN; Bulimia Nervosa; Obesity
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia Nervosa; Feeding and Eating Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HAPIFED (Experimental): HAPIFED therapy
  Interventions: Behavioral: HAPIFED
- CBT-E (Active Comparator): CBT-E therapy
  Interventions: Behavioral: CBT-E

INTERVENTIONS:
Behavioral: HAPIFED — HAPIFED is adapted from CBT to promote a positive relationship with food, eating and activity, appetite awareness, and weight loss to be achieved over a longer and more intensive period of therapy, thus recognizing the importance of longer-term therapy in weight loss (Casazza et al., 2013). Notably, HAPIFED is also multidisciplinary. Clinical practice and consensus views are to utilize the special expertise of dietitians and other allied health professionals (Robinson, 2009).
  Arms: HAPIFED
Behavioral: CBT-E — CBT-E therapy
  Arms: CBT-E

SUMMARY:
The investigators have developed a new integrated therapy, namely a Healthy Approach to weIght management and Food in Eating Disorders (HAPIFED). HAPIFED is an enhanced behavioral weight loss therapy integrated with CBT for the management of EDs. HAPIFED uses CBT to treat ED behaviors and body image distress, whilst simultaneously emphasize a healthy lifestyle, the role of food and physical activity in mood regulation, and revised but clinically meaningful goals for weight loss. The investigators propose a randomized controlled trial (RCT) that will compare HAPIFED to CBT-E in people with obesity and either BN or BED. The two main aims will be to reduce symptoms of ED and to improve weight management. The RCT will be conducted in Sydney and in São Paulo with a one year follow-up.

DETAILED DESCRIPTION:
In sum, a new approach in management of the increasing numbers of obese people with BN and BED is needed. The investigators propose a RCT that will compare a novel therapy HAPIFED with the current 'gold-standard' trans diagnostic treatment, CBT-E. HAPIFED has been developed by the CIs and is based on recent developments in psychological approaches to obesity in general (as highlighted in Casazza et al.'s (2013) paper on "Myths, presumptions and facts about obesity") and in people with co-morbid obesity and BN or BED. Unlike CBT-E, it allows reduced energy intake and education around specific food choices - a necessary element in weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of threshold or subthreshold for Bulimia Nervosa or Binge Eating Disorder (DSM-5/ICD-11)
* BMI between ≥ 27 and < 40

Exclusion Criteria:

* Diagnosis of psychosis, bipolar disorder or substance abuse dependence and/or a high level of suicide risk.
* Use of weight loss medication or medications that interfere with appetite.
* Cushing or Prader-Willi syndromes
* History of bariatric surgery
* Patients who are already in treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Sustained change weight (for less) of 5% of previous body weight. This is a level known to improve physical health (metabolic) outcomes. | Baseline, 25-weeks (end) treatment, 6 and12 months follow-up.
  Change of 5% of body weight.

SECONDARY OUTCOMES:
Change in binge eating frequency | Baseline, 14 weeks (mid) treatment, and 25 weeks (end) treatment, 6 and 12 months follow-up.
  Change (for less) in binge eating frequency as measured on the Eating Disorder Examintaion Questionnaire
Severity of loss of control over eating | Baseline, 14 weeks (mid) treatment, and 25 weeks (end) treatment, 6 and 12 months follow-up.
  Change (for less) in the Global (total) Loss of Control over Eating Scale (LOCES) score
Change in severity of binge eating | Baseline, 14 weeks (mid) treatment, and 25 weeks (end) treatment, 6 and 12 months follow-up.
  Binge eating severity as measured by a reduced total score on the Binge Eating Scale questionnaire
Improved metabolic indicators of weight management | Baseline, 25 weeks (end) treatment
  Waist and Hip circumference and blood markers (Blood fasting lipid profile, fasting glucose matched with insulin, liver function tests, electrolytes, urea, uric acid and creatinine.
Change in the levels of depression, anxiety and stress. | Baseline, 14 weeks (mid) treatment, and 25 weeks (end) treatment, 6 and 12 months follow-up.
  Changed level of depression, anxiety and stress as measured on the Depression, Anxiety and Stress Scale 21 item questionnaire - subscale scores of depression, anxiety and stress
Health related quality of life | Baseline, 14 weeks (mid) treatment, and 25 weeks (end) treatment, 6 and 12 months follow-up.
  Improved physical and mental health related quality of life as measured by increased scores on the Short Form 12-item survey (SF-12) Physical and Mental Health Component scores

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Claudino, MD, Ph.D, Principal Investigator — Federal University of São Paulo
Locations (1):
- Universidade Federal de Sao Paulo (UNIFESP), São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Palavras MA, Hay P, Filho CA, Claudino A. The Efficacy of Psychological Therapies in Reducing Weight and Binge Eating in People with Bulimia Nervosa and Binge Eating Disorder Who Are Overweight or Obese-A Critical Synthesis and Meta-Analyses. Nutrients. 2017 Mar 17;9(3):299. doi: 10.3390/nu9030299. PMID 28304341
- [Background] Palavras MA, Hay P, Touyz S, Sainsbury A, da Luz F, Swinbourne J, Estella NM, Claudino A. Comparing cognitive behavioural therapy for eating disorders integrated with behavioural weight loss therapy to cognitive behavioural therapy-enhanced alone in overweight or obese people with bulimia nervosa or binge eating disorder: study protocol for a randomised controlled trial. Trials. 2015 Dec 18;16:578. doi: 10.1186/s13063-015-1079-1. PMID 26683478
- [Background] Palavras MA, Hay P, Claudino A. An Investigation of the Clinical Utility of the Proposed ICD-11 and DSM-5 Diagnostic Schemes for Eating Disorders Characterized by Recurrent Binge Eating in People with a High BMI. Nutrients. 2018 Nov 13;10(11):1751. doi: 10.3390/nu10111751. PMID 30428611
- [Derived] Hay P, Palavras MA, da Luz FQ, Dos Anjos Garnes S, Sainsbury A, Touyz S, Appolinario JC, Claudino AM. Physical and mental health outcomes of an integrated cognitive behavioural and weight management therapy for people with an eating disorder characterized by binge eating and a high body mass index: a randomized controlled trial. BMC Psychiatry. 2022 May 24;22(1):355. doi: 10.1186/s12888-022-04005-y. PMID 35610603
- [Derived] Palavras MA, Hay P, Mannan H, da Luz FQ, Sainsbury A, Touyz S, Claudino AM. Integrated weight loss and cognitive behavioural therapy (CBT) for the treatment of recurrent binge eating and high body mass index: a randomized controlled trial. Eat Weight Disord. 2021 Feb;26(1):249-262. doi: 10.1007/s40519-020-00846-2. Epub 2020 Jan 25. PMID 31983019